CLINICAL TRIAL: NCT07103863
Title: A Prospective Study on the Prognostic Assessment of Light Chain Type Cardiac Amyloidosis (AL-CA) Based on Multimodal Fusion Radiomics Model of 18F-FAPI PET/CT and 3D CMR
Brief Title: Multimodal Radiomics Model (18F-FAPI PET/CT + CMR) for AL Cardiac Amyloidosis Prognosis
Acronym: AL-CA
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingAnzhen dongwei; High Level research funding (Other Grant/Funding Number: Beijing Anzhen Hospital)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-02

CONDITIONS: AL Amyloidosis (AL); Cardiac Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rationale: AL-CA: Clearly identifies the disease population (Light-chain Cardiac Amyloidosis). Mul

SUMMARY:
1. Goal of the Study:

   The goal of this prospective observational study is to develop and validate a novel, non-invasive method for predicting the prognosis of patients with light-chain cardiac amyloidosis (AL-CA). This method integrates advanced multi-modal imaging techniques and artificial intelligence (radiomics) to provide early and accurate assessment of treatment response and survival outcomes.
2. Main Question:

   Can a multi-modal radiomics model, based on the fusion of [¹⁸F]FAPI PET/CT (assessing fibroblast activation) and 3D Cardiac MRI (CMR) (assessing structural damage) imaging data, accurately predict 12-month all-cause mortality and dynamically track disease progression in patients with AL-CA receiving standard care?
3. Participants:

   Population: Patients diagnosed with AL-CA (confirmed by endomyocardial biopsy or extracardiac biopsy plus specific cardiac criteria: NT-proBNP >332 pg/mL, mean left ventricular wall thickness >12 mm, excluding hypertension/other causes).

   Setting: Single-center study at Beijing Anzhen Hospital, Capital Medical University.

   Number: 49 patients (calculated sample size accounting for dropouts).

   Key Criteria:

   Inclusion: Confirmed AL-CA diagnosis, receiving standard AL-CA treatment (chemotherapy e.g., Daratumumab-based regimen + supportive cardiac care).

   Exclusion: Active infection, advanced malignancy (life expectancy <12 months), severe cognitive impairment/immobility affecting imaging compliance/follow-up.
4. Study Design & Procedures:

   Design: Single-center prospective cohort study.

   Intervention: Participants receive standard-of-care treatment for AL-CA as per guidelines (chemotherapy regimen based on Daratumumab, Bortezomib, Cyclophosphamide, Dexamethasone; tailored cardiac support including diuretics, rate control, anticoagulation if needed).

   Procedures:

   Baseline: Upon enrollment, participants undergo comprehensive assessment: [¹⁸F]FAPI PET/CT scan, 3D CMR scan, blood tests (NT-proBNP, troponin, free light chains, etc.), clinical staging (Mayo 2012), functional assessment (NYHA class), quality of life questionnaire (KCCQ).

   Imaging: Specialized software (Siemens True D) performs cross-platform fusion of PET/CT and 3D CMR images. Radiomics features are extracted from the fused images using dedicated software (Siemens FeAture Explorer).

   Follow-up:

   Clinical: Every 3 months (symptoms, medication adherence, adverse events, lab tests including NT-proBNP).

   Imaging: Repeat [¹⁸F]FAPI PET/CT and 3D CMR scans at 6 months post-baseline. Radiomics features are extracted again.

   Endpoints: Primary endpoint is 12-month all-cause mortality. Secondary endpoints include re-hospitalization rates and changes in NYHA class. Follow-up continues until the 12-month endpoint for all participants.

   Data Analysis: Machine learning (LASSO-Cox regression) is used to select key radiomics features from baseline and 6-month scans and integrate them with quantitative imaging parameters (FAPI uptake volume, SUVmax, LGE burden, ECV) and clinical data to build prognostic models predicting 12-month survival.
5. Comparison:

Researchers will compare the predictive performance of the developed multi-modal radiomics model against:

* Traditional clinical biomarkers: NT-proBNP levels and Mayo Clinic staging.
* Standard quantitative imaging parameters alone: Such as myocardial FAPI uptake volume, SUVmax, or CMR-derived extracellular volume (ECV) measured at baseline and 6 months.

The goal is to demonstrate superior accuracy in predicting 12-month all-cause mortality using the integrated radiomics approach.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed AL cardiac amyloidosis (AL-CA) by endocardial biopsy;
* Pathologically confirmed AL-CA by extracardiac (bone marrow, adipose tissue, tongue muscle, etc.) biopsy, with serum N-terminal pro-brain natriuretic peptide (NT-proBNP) > 332 pg/mL, left ventricular mean wall thickness > 12 mm, and exclusion of hypertension and other secondary causes of left ventricular hypertrophy;
* Receiving standard AL-CA treatment regimens (including chemotherapy and supportive therapy).

Exclusion Criteria:

* Complicated with active infection or advanced malignant tumor (expected survival time < 12 months);
* Presence of severe cognitive impairment, limited mobility, or other conditions that affect compliance with imaging examinations or the completeness of follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Design
  1. Study Type: Single-center prospective cohort study (evaluating the prognostic value of radiomics parameters under standardized treatment).
  2. Study Population: Patients with suspected or confirmed cardiac light-chain amyloidosis (AL-CA) via endocardial or extracardiac biopsy who are admitted to the Department of Hematology, Beijing Anzhen Hospital, from Feburary 2025 to August 2028.
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
12-month survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: wei dong, MD,PHD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No